CLINICAL TRIAL: NCT07202611
Title: In Vitro Culture of Autologous Dendritic and Natural Killer Cells for the Treatment of Patients With Non-small Cell Lung Cancer
Brief Title: DC/NK Cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Clinical Trial Center (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, Clinical Associate Professor, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201904109MIFC
Record Dates: First submitted 2025-01-07; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (NSCLC)
Keywords: lung cancer; cell therapy; NK cell; Dendritic cell
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Patients who diagnosed as histologically or cytologically with stage IIIB or stage IV non-small cell lung cancer (NSCLC) or patients with recurrence or progression following multimodal treatments (radiotherapy, surgical resection, or therapeutic chemoradiotherapy for locally advanced disease), and have undergone at least two systemic therapies for advanced NSCLC, including platinum-based chemotherapy, anti-PD-1 therapy, and/or other targeted therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- In vitro culture of autologous dendritic and natural killer cells for the treatment of patients with (Experimental)
  Interventions: Biological: In vitro culture of autologous dendritic and natural killer cells for the treatment of patients with non-small cell lung cancer

INTERVENTIONS:
Biological: In vitro culture of autologous dendritic and natural killer cells for the treatment of patients with non-small cell lung cancer — The primary objective of this trial is to test the safety of formulations containing dendritic cells (DCs) and natural killer (NK) cells cultured in vitro. By evaluating the reactions following the administration of autologous dendritic cells via axillary lymph node injection and natural killer cells via intravenous injection, the study aims to determine the safety profile of these trial products for human use.

SUMMARY:
Primary Outcomes The primary objective of this trial is to test the safety of formulations containing dendritic cells (DCs) and natural killer (NK) cells cultured in vitro. By evaluating the reactions following the administration of autologous dendritic cells via axillary lymph node injection and natural killer cells via intravenous injection, the study aims to determine the safety profile of these trial products for human use.

Secondary Outcomes

To verify the success rate of the cultured cell formulations and assess the cytotoxic capacity of natural killer cells in targeting and killing tumor cells. The evaluation of these secondary objectives involves analyzing specific subcategories, which can be divided into two major components:

1. Validation of Cultured Cell Preparation Success: Assessing the proliferation rate, recovery rate, survival rate, and tumor-killing capacity of the cultured autologous dendritic cells and natural killer cells.
2. Validation of Antitumor Effectiveness: Evaluating the antitumor efficacy of the trial products administered via axillary lymph node injection of autologous dendritic cells and intravenous infusion of autologous natural killer cells.

DETAILED DESCRIPTION:
Research Background and Current Status of Medical Technology According to data from the Ministry of Health, cancer has consistently ranked as the leading cause of death in Taiwan. Although various treatments for cancer, including surgery, chemotherapy, and radiotherapy, are currently available, there is still significant room for improvement in terms of extending survival and reducing side effects. Recently, research on natural killer (NK) cell therapy has gained attention both domestically and internationally. While the therapeutic effects remain uncertain and most countries are still in the clinical trial stage, preliminary results and studies from other countries suggest that combining NK cell therapy with traditional treatments like chemotherapy or radiotherapy may provide additional benefits for cancer patients.

Natural killer cells are among the first-line innate immune defenses in the human body and are considered one of the most potent and effective cells for combating cancer and viral infections. Compared to other anti-cancer immune cells, such as cytotoxic T cells or dendritic cells, NK cells exhibit stronger cytotoxicity, a broader spectrum of activity, and are not restricted by tissue compatibility antigens. They can directly attack cancer cells without the need for prior sensitization. Since the discovery of NK cells in the 1970s, immunologists have hypothesized that expanding NK cells in large quantities and reinfusing them into patients could achieve anti-cancer effects, enhance immune regulation, and improve overall immunity. This forms the theoretical basis of NK cell therapy.

In simple terms, NK cell therapy involves the use of cell culture techniques to rapidly proliferate a patient's NK cells in vitro and then reinject them into the patient. This approach aims to boost the patient's innate anti-cancer capacity and support conventional therapies in achieving cancer treatment goals.

Laboratory studies using animal models and in vitro experiments have highlighted several theoretical advantages of NK cell therapy for cancer treatment:

1. NK cells exhibit the strongest anti-cancer activity in the human body, directly killing cancer cells and inhibiting tumor growth and spread.
2. NK cells suppress the formation of new blood vessels around tumors, restricting the supply of nutrients necessary for tumor growth.

Although the clinical effectiveness of NK cell therapy for cancer in humans has yet to be confirmed, some preliminary international studies suggest that adding activated NK cells or cytokine-induced killer (CIK) cells to standard treatments may help inhibit the spread of cancer cells and slow disease progression.

Characteristics of Human Cell Therapy Products and Usage Experience

1. Cell Source and Characteristics Source: Autologous cells

   Characteristics:

   Dendritic cells (DCs) have the ability to activate adaptive immune functions. NK cells possess tumor-killing capabilities.

   Rationale for Use in This Indication:

   Preliminary clinical studies indicate that in non-small cell lung cancer (NSCLC) patients, groups receiving NK cell (or NK + DC) immunotherapy in addition to traditional treatments (surgery, chemotherapy, or radiotherapy) showed better outcomes in individual trials compared to control groups that received only traditional treatments. These outcomes included improved objective response rates (ORR), progression-free survival (PFS), overall survival (OS), and, in some cases, enhanced quality of life (refer to the summary table on the next page for details).
2. Usage Experience Numerous clinical trials have already been conducted internationally. The investigational drug in this trial is being tested in humans for the first time.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility of Participants:

   o Diagnosed histologically or cytologically with stage IIIB or stage IV non-small cell lung cancer (NSCLC) or patients with recurrence or progression following multimodal treatments (radiotherapy, surgical resection, or therapeutic chemoradiotherapy for locally advanced disease).
   * Have undergone at least two systemic therapies for advanced NSCLC, including platinum-based chemotherapy, anti-PD-1 therapy, and/or other targeted therapies.
2. At Least One Measurable Lesion:

   o The measurable lesion must not undergo radiotherapy during the cell therapy period.
3. Age:

   o ≥20 years.
4. Weight:

   o Between 40 and 100 kg.
5. Normal Blood Count (based on test results within 4 weeks before blood collection for cell preparation):

   o White blood cells (WBC): ≥3000/mm³.

   o Lymphocytes: ≥1000/mm³.
   * Hemoglobin: ≥10 g/dL.
   * Platelets: ≥100,000/mm³.
6. Normal Liver and Kidney Function (based on test results within 4 weeks before blood collection for cell preparation):

   * Creatinine: ≤1.25× the upper limit of normal (ULN).
   * Total bilirubin: ≤1.5× ULN.
   * SGOT (AST): ≤3× ULN.
   * SGPT (ALT): ≤3× ULN.
7. Informed Consent:

   o Participants must sign the consent form.
8. ECOG Performance Status:

   o Score of 0-1.
9. For Women of Childbearing Age:

   * Must agree to use effective contraception during the trial.

Exclusion Criteria:

1. Positive Test Results for the Following Infections:

   o HCV (HCV antibody-positive).
   * HBV (HBsAg-positive).
   * HIV (HIV antibody-positive).
   * HTLV (HTLV antibody-positive).
   * Syphilis (Treponema pallidum antibody-positive).
   * Tuberculosis (TB culture-positive).
2. ECOG Performance Status:

   o Score of 2-4.
3. Albumin Intolerance:

   o Participants who cannot tolerate albumin.
4. Short Life Expectancy:

   o Life expectancy estimated by the physician to be less than 12 weeks.
5. Participation in Other Clinical Trials:

   o Within 30 days prior to entering this trial.
6. Pregnancy or Breastfeeding:

   o Positive pregnancy test or currently breastfeeding.
7. Other Medical Conditions:

   o Immunodeficiency, severe heart or lung dysfunction, coagulation disorders, unresolved side effects from prior cancer therapy (not recovered to CTCAE grade 1), prior transplant surgery, or deemed unsuitable by the physician.
8. Noncompliance:

   o Unable to adhere to follow-up or examination procedures.
9. Concurrent Cancer:

   o Other cancers diagnosed within the past 2 years.
10. Specific Complications:

    * Brain metastases, leptomeningeal disease, or spinal cord compression.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events Following Administration of Autologous Dendritic Cells (via Axillary Lymph Node Injection) and Natural Killer Cells (via Intravenous Injection) cultured in vitro | 12 weeks
  The primary objective of this trial is to evaluate the safety profile of in vitro-cultured dendritic cells (DCs) and natural killer (NK) cells. Specifically, the study will assess adverse reactions, including incidence, type, and severity of treatment-emergent adverse events, following administration of autologous DCs via axillary lymph node injection and NK cells via intravenous injection.

SECONDARY OUTCOMES:
Number of Participants with Successful Cultured Cell Preparation (Defined by ≥80% Cell Viability and Absence of Contamination) | 12 weeks
  Validation will be based on cell viability, sterility testing, and phenotypic confirmation. A successful preparation is defined as viability ≥80%, absence of bacterial/mycoplasma contamination, and retention of lineage-specific surface markers as assessed by flow cytometry.
Validation of Antitumor Effectiveness (In Vitro) | 12 weeks
  Percentage of Tumor Cells Exhibiting Reduced Viability After Treatment (MTT Assay)
Proportion of Participants with Tumor Response (Complete Response, Partial Response, or Stable Disease per RECIST v1.1) | 12 weeks
  Number of Participants with Treatment-Emergent Objective Tumor Regression (≥30% Reduction in Target Lesions per RECIST v1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Huwei, YUNLIN, Taiwan

IPD SHARING:
Plan to Share IPD: No